CLINICAL TRIAL: NCT00250055
Title: Non-Invasive, Real-time Technology for Diagnosis of Cervical Tissue
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This is not Clinical Trial and was inadvertently entered in this system.
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1104C
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cervix; Cancer
Keywords: NIH; Non-Invasive diagnosis of cervical tissue; Los Alamos/NIH
MeSH Terms: conditions — Neoplasms | interventions — Colposcopy; Spectrum Analysis; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Colposcopy, Spectroscopy, and Biopsy — During the colposcopy or LEEP (Loop Electrical Excision Procedure) procedure, or during pelvic exams before surgery after the doctor applies 3% acetic acid to the cervix, the doctor then positions the colposcope to take pictures of the patient's cervix. Digital pictures are taken of the patient's cervix under white light using a colposcopy imaging system. These pictures are annotated by the doctor during the appointment to mark the spectroscopy sites.

SUMMARY:
In general, to determine the sensitivity of light transport to tissue from morphological features of clinical significance.

Determine how specific structural features contribute to light scattering. Investigate light scattering differences in tumorigenic and nontumorigenic cells.

Develop and implement quantitative and sensitive methods for measuring morphological properties.

Clinical measurements.

DETAILED DESCRIPTION:
Patients undergoing a colposcopy will also have spectroscopy measurements taken and an extra biopsy of suspicious tissue.

ELIGIBILITY:
Inclusion Criteria:

* Patients with abnormal Pap smears who are referred for colposcopy.

Exclusion criteria include:

* Anyone of the male sex since this study focuses on cervical cell abnormalities
* Any woman who has had a hysterectomy, LEEP, or chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2004-04 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
The objective of this study is to determine whether non-invasive measurements of light transport through tissue can identify pre-cancerous and cancerous conditions. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Smith, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States